CLINICAL TRIAL: NCT06156228
Title: Multilevel Intervention of COVID-19 Vaccine Uptake Among Latinos
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant funding was terminated.
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HS-2022-0096
Record Dates: First submitted 2023-11-30; First posted 2023-12-05 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Vaccine Hesitancy
Keywords: Vaccine Promotion
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Investigators will implement a multilevel intervention in 10 clinics that will be randomized to either a Standard Clinical Practice consisting of standard clinic-based strategies to promote vaccine uptake among patients or a Multilevel Intervention consisting of an individualized/tailored intervention delivered by Health Educators working within the clinics plus a multi-component community intervention delivered by community promotores.
Who Masked: Participant, Care Provider, Investigator
Masking Description: In order to generate evidence that reflects real-world circumstances and is generalizable to a broad patient population served by Federally Qualified Health Centers, Investigators will evaluate our proposed intervention in a single-blind, pragmatic, cluster randomized trial, whereby 10 clinics will be randomized at a ratio of 1:1 to one of two conditions. The first being standard clinical practice and the second being the intervention which will include motivational interviews where health educators can assist with scheduling their vaccine appointments should the clinic patient opt for that. The study participants will not know whether they are placed on the intervention or control group and their care providers will also be unaware. This will ensure balance across study conditions regarding clinic patient characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multilevel Intervention (Experimental): The Multilevel Intervention condition will receive tailored and targeted messages about vaccination. Health educators will also deliver motivational interview sessions to patients eligible to receive the vaccines during the first 6 months of the study. To supplement these encounters, health educators will also send patients mail, emails and/or text message-based informational materials (including videos, testimonials, and resources) that reinforce the benfits of vaccines.
  Interventions: Behavioral: Multilevel Intervention
- Standard Clinical Practice (No Intervention): Standard clinical practice consisting of generic patient outreach to promote vaccine uptake among Latino patients.

INTERVENTIONS:
Behavioral: Multilevel Intervention — Clinic patients from the randomly assigned intervention clinics will be provided with additional vaccine information and will have the opportunity to ask any questions they might have about any of the 4 study focused vaccines (COVID-19, Shingles, Pneumococcal, Influenza). Health educators will provide them with additional information, address any misinformation and disinformation and will offer to schedule their vaccine appointment(s) for them.
  Arms: Multilevel Intervention

SUMMARY:
This study is significant as it targets a population that has exceptionally high rates of morbidity and mortality due to COVID-19, influenza, pneumococcal pneumonia and shingles; and who demonstrate significant mistrust towards the vaccines. It is innovative in that investigators will harness the research team's extensive experience in developing multi-level and tailored interventions working with community partners to increase adult vaccine uptake among Latinos. Through this project the investigators will develop the experience and infrastructure for a scalable community-academic model that can be deployed and adapted to other communities (especially those with prevalent vaccine resistance) and other emerging public health threats. There is great potential for short- and long-term public health/economic impact in increasing adult vaccine uptake among high risk populations such as Latinos. This work will contribute to the body of evidence for effective behavioral- and community-based strategies to improve the health of Latinos.

DETAILED DESCRIPTION:
COVID-19 disparities are central to its local and national spread. Since the emergence of the novel coronavirus (SARS-CoV-2), there have been over 104.8 million confirmed cases worldwide, with the U.S. leading in number cases and deaths (as of this writing, >26.6 mil and 455K+, respectively)1 and California leading the U.S. with >3.3 mil cases.1 COVID-19 (the disease caused by SARS-CoV-2) is spread primarily from person-to-person through close and sustained contact with an infected individual. Unfortunately, the U.S. response to the pandemic has largely been left to state and local governments, which has resulted in mixed results. Ethnic/racial minority individuals are at an increased risk of acquiring SARS-CoV-2 infection compared to Whites, and demonstrate worse clinical outcomes from COVID-19. For example, Latinos experience a 2.5 times higher death rate from COVID-19 compared to Whites.2 In California, Latinos account for the highest percent of COVID-19 cases (55%) and deaths (46%) despite similar population percentages as Whites (38.9% vs. 36.6%, respectively).3 In San Diego County, Latinos have the highest case rates (56.3%) compared to any other ethnic group.4 These data show profound and clear disparities affecting Latinos in California and San Diego County.

Determinants of COVID-19 disparities among Latinos are the result of pervasive systemic socioeconomic disparities. Latinos are disproportionately represented in occupations deemed as 'essential' (78%)5 and suffer from high rates of poverty (18.3%) compared to Whites (59% and 8.7%, respectively).6 Together, these factors place Latinos at a greater need to continue working outside the home, thereby increasing risk of exposure to SARS-CoV-2. In addition, due to both economic and cultural factors, Latinos may live in smaller housing units with multi-generational households which makes practicing social distancing dificult.7 Latinos also have higher rates of obesity, hypertension and type 2 diabetes; all of which are known risk factors for severe COVID-19 complications.8 Lastly, due to educational disparities and historical distrust of government entities,9 Latinos may be more vulnerable to misinformation regarding COVID-19, and thus not adopt or adhere to preventive recommendations.10 These disparities highlight the urgent need to reduce the COVID-19 burden among Latinos.

Vaccine hesitancy and mistrust among Latinos can further exacerbate the burden of COVID-19 experienced by this group. To date, the national response to the COVID-19 pandemic and subsequent vaccination rollout has been largely inadequate. Common cited concerns of the COVID-19 vaccine include the speed at which they were developed and approved, the newness of the mRNA-based technology (Moderna & Pfizer), the relatively short-term efficacy and safety data available, and the risk of potential side effects. To compound these concerns, social media and other platforms (e.g., Facebook & YouTube) have been used to propagate misinformation regarding COVID-19 and the COVID-19 vaccines. These factors, in combination, have degraded the trust of Latinos for the COVID-19 vaccine. Thus, it is clear that Latinos are a priority group to implement strategies to increase trust in the COVID-19 vaccine and increase COVID-19 vaccine uptake. FHCSD provides an ideal setting to conduct research centered on establishing effective methods for reaching and serving large numbers of Latinos.

More recently, it has become apparent that COVID-19 vaccination will be a yearly and seasonal vaccine, similar to influenza. Given this, it is important to leverage vaccination efforts and communication campaigns that target multiple vaccines. These include: COVID-19, influenza, pneumococcal pneumonia and shingles. Evidence indicates that similar ethnic disparities exist for flu (11), pneumococcal pneumonia (12), and shingles (13).

ELIGIBILITY:
Inclusion Criteria:

* Be a patient of an intervention participating clinic
* Be an adult 18+
* Self identify as Latino

Exclusion Criteria:

* Be planning to move out of San Diego County in the next 2 years
* Have cognitive impairment making them unable to complete informed consent
* Have any contraindications to receiving the 4 study vaccines (COVID-19, Pneumococcal, Shingles, Influenza)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Vaccination of Latino clinic patients | 1 year
  Test Multilevel Intervention effectiveness at baseline, 6-months & 12-months on Latino patient's vaccine uptake for COVID-19, Pneumococcal, Shingles and Influenza vs. Latino patients receiving Standard Clinical Practice.

SECONDARY OUTCOMES:
Psychosocial and Individual-level outcomes | 1 year
  Test longer-term (24-mo) effectiveness of the Multilevel Intervention on psychosocial & quality of life outcomes among a subgroup of 200 Latino clinic patients.

OTHER OUTCOMES:
Implementation Assessment | 1 year
  Assess implementation process & fidelity, including intervention acceptability & perceived feasibility by patients, clinic staff, community agencies and stakeholders at baseline, 3 month, 6 month and 12 month timepoints.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Family Health Centers San Diego, San Diego, California
  - San Diego State University Research Foundation, San Diego, California